CLINICAL TRIAL: NCT05807958
Title: Validation of the Benefit of Allergy Testing of Soldiers Prepared for International Mission with Specific Allergen Panels
Brief Title: Allergy Testing of Soldiers Prepared for International Mission
Acronym: SPAT_ABL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Astrid Military Hospital (Other)
Responsible Party: Principal Investigator, Ilan Baron, Medical doctor, Queen Astrid Military Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22467
Record Dates: First submitted 2023-03-14; First posted 2023-04-11 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Adult Military Personnel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Skin Prick Automated Test (Experimental)
  Interventions: Device: Skin Prick Automated Test

INTERVENTIONS:
Device: Skin Prick Automated Test — A skin prick automated test will be performed in each participant.

SUMMARY:
The goal of this prospective mono centric study is to identify relevant commercially available allergen extracts for allergy testing in soldiers prepared for international mission.

Participants will receive a skin prick test with the skin prick automated test device including 22 allergens and 2 controls on both forearms.

ELIGIBILITY:
Inclusion Criteria:

* Adult military personnel (18-65y) will be included. Soldiers with and without previous exposure to allergens in the regions of interest will be included. Soldiers who are performing desk tasks and not selected for international missions will serve as controls.

Exclusion Criteria:

* Skin pathology like chronic or exuberant urticaria, dermographism, chronic dermatitis that needs daily treatment
* Use of antihistaminic medication < 7 days before the start of the study
* Use of tricyclic antidepressants (antihistamine activity) < 7 days before the start of the study
* Use of topical corticoids on the forearm < 7 days before the start of the study
* Use of Omalizumab < 6 months before the start of the study
* Pregnancy: there is a remote possibility of inducing a systemic allergic reaction that could induce uterine contractions or necessitate the use of epinephrine (thought to cause constriction of the umbilical artery).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
Allergens with positive skin reaction | baseline
  Positive skin reactions of top ranked allergens required to identify 95% of sensitised individuals

SECONDARY OUTCOMES:
Self-reported allergic diseases | baseline
  Percentage of soldiers with self-reported allergic diseases derived from questionnaire
Work Performance & Activity Impairment | baseline
  Total score of Work Performance & Activity Impairment questionnaire, 0-100%, higher score means worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Baron, MD, Principal Investigator — Military Hospital Queen Astrid
Locations (1):
- Military Hospital Queen Astrid, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gorris S, Uyttebroek S, Backaert W, Jorissen M, Schrijvers R, Thompson MJ, Loeckx D, Seys SF, Van Gerven L, Hellings PW. Reduced intra-subject variability of an automated skin prick test device compared to a manual test. Allergy. 2023 May;78(5):1366-1368. doi: 10.1111/all.15619. Epub 2022 Dec 26. No abstract available. PMID 36495473
- [Derived] Gorris S, Baron I, De Brouwer J, Vanden Daele A, Verstraelen J, Loeckx D, Bousquet J, Van Gerven L, Seys SF. Sensitisation patterns and burden of uncontrolled respiratory allergy symptoms in military personnel. BMJ Mil Health. 2025 Jun 25:military-2025-003006. doi: 10.1136/military-2025-003006. Online ahead of print. PMID 40562451